CLINICAL TRIAL: NCT00637715
Title: Evaluation of the Effect of 10 mg Alfuzosin (Alfetim Uno®) o. d. in Patients Presenting Low-Urinary Tract Symptoms
Brief Title: Once Daily Given Alfuzosin in the Treatment of BPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8758
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alfuzosin

SUMMARY:
Collection of the data on the safety and efficacy of the once daily administration of the alfuzosin preparation /Alfetim Uno® l0 mg/ at patients with lower urinary tract symptoms/complaints rendering possible the presence of benign prostatic hyperplasia, in the course of everyday practice

ELIGIBILITY:
Inclusion Criteria:

* Sexually active male patient with lower urinary tract symptoms indicative of severe BPH, at whom disturbances of urinary retention and urination are present

Exclusion Criteria:

* Necessity of surgical intervention immediately or within 12 months because of BPH
* The patient has earlier /within 6 months/ obtained treatment because of BPH
* The patient did not improve on earlier alpha-1 blocker treatment
* Known hypersensitivity to alfuzosin
* Orthostatic hypotension in the history
* Concomitant application with another alpha-1 blocker
* Hepatic insufficiency /AST, ALT 3 fold of the upper limit of the normal value/
* Severe renal insufficiency /se creatinine greater than or equal to 150 umol/l/
* Intestinal obstruction /because of the castor oil content of the drug/
* Tumorous disease
* Severe, life threatening state

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-10; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To collect additional clinical data on the safety profile and efficacy of alfuzosin 10 mg o. d. in patients with low-urinary tract symptoms caused by benign prostatic hyperplasia (BPH) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Eros, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Budapest, Hungary